CLINICAL TRIAL: NCT02685943
Title: "Collaborative Assessment and Management of Suicidality" (CAMS) in Comparison to "Treatment as Usual" (TAU) for Suicidal Patients: a Randomized Controlled Trial
Brief Title: A Randomized Trial for Suicidal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: The Catholic University of America (Other); Helse Sor-Ost (Other Government); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 2014/465
Record Dates: First submitted 2016-02-08; First posted 2016-02-19 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Suicidal Ideation; Attempted Suicide; Suicide
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAMS treatment (Experimental): Psychotherapy using the Collaborative Assessment and Management of Suicidality framework
  Interventions: Behavioral: Psychotherapy
- Treatment as usual (Active Comparator): Ordinary treatment for suicidal patients
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy

SUMMARY:
Although suicide risk is highly prevalent among the patient population in mental health care, remarkably little research exists on effective treatments. Among a small set of novel approaches, CAMS is particularly promising. The investigators compare CAMS to TAU in a randomized controlled trial at four departments in Vestre Viken Hospital Trust, hypothesizing CAMS to be the superior approach. Primary outcome measures are suicidal ideation and suicide attempts, with secondary outcome measures including general symptoms of mental health problems. Changes in the outcome measures are compared between the two groups from baseline to 6 and 12 months after patients are included in the study. The study has the potential to impact the science of treating suicidal individuals and it could benefit the general public by establishing CAMS as an effective clinical approach for rapidly reducing suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* Significant suicide ideation on Beck's Scale for Suicide Ideation (score 13 and above). Informed consent to participate.

Exclusion Criteria:

* Active psychosis, cognitive or physical impairment or other problems that preclude the ability to understand the study procedures and provide informed consent, non-Norwegian speaking subjects

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in scores on Beck's Scale for Suicide Ideation (BSSI) | From baseline to 6 and 12 months after patient is included in the study
  Interview scale with 19 items that measures a patient's suicidal ideation at its worst point in the past 2 weeks.

SECONDARY OUTCOMES:
Changes in scores on The Outcome Questionaire 45 (OQ-45) | From baseline to 6 and 12 months after patient is included in the study
  A 45-item questionnaire designed to measure key areas of mental health functioning (symptoms, interpersonal problems and social role functioning)
Norwegian Patient Registry (NPR) data | Yearly for five years after study inclusion
  Data entered in the NPR on self harm, suicide attempts, new hospital admissions to health treatments, discharge diagnosis, intoxication, and death by any causes.
Changes in scores on Suicide Attempt Self-Injury Count (SASI-C) | changes from baseline to 6 and 12 months after patient is included in the study
  An interview covering past self-inflicted injuries and categorizing them into suicide attempts and non-suicidal acts. The tool also creates counts of self-inflicted injuries by method, medical risk severity and lethality

CONTACTS AND LOCATIONS:
Overall Officials: Roar Fosse, Ph.D., Principal Investigator — Division of mental health and addiction, Vestre Viken
Locations (1):
- Vestre Viken Helseforetak, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared/ published

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Ryberg W, Fosse R, Zahl PH, Brorson I, Moller P, Landro NI, Jobes D. Collaborative Assessment and Management of Suicidality (CAMS) compared to treatment as usual (TAU) for suicidal patients: study protocol for a randomized controlled trial. Trials. 2016 Oct 3;17(1):481. doi: 10.1186/s13063-016-1602-z. PMID 27716298